CLINICAL TRIAL: NCT05224414
Title: Interpretation Bias as a Mechanism of Treatment Response in OCD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Martha J Falkenstein, Director of Research, OCD Institute, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2022P000190
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive bias modification with treatment as usual (Experimental): Participants in this group will receive usual treatment in the program up to 12 sessions of a digital cognitive training targeting interpretation bias
  Interventions: Behavioral: Cognitive bias modification for interpretation bias
- Psychoeducation with treatment as usual (Sham Comparator): Participants in this group will receive usual treatment in the program up to 12 sessions of digitized psychoeducation
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Cognitive bias modification for interpretation bias — Sessions of scenario-based CBM-I training for OCD will be administered, based on the widely-used paradigm of ambiguous scenario training developed by Mathews and Mackintosh (2000), in which participants are presented with scenarios that are ambiguous in whether or not they are threatening. Participants will complete a computer task consisting of a series of written scenarios designed to improve interpretation and attributional biases; these scenarios conclude with word fragments, which participants must fill in to resolve the ambiguity.
  Arms: Cognitive bias modification with treatment as usual
Behavioral: Psychoeducation — Sessions of psychoeducation will be administered, which will describe symptoms of anxiety, the nature of biased thinking in anxiety, and summarize common psychosocial as well as pharmacological treatments for anxiety. The sessions will provide relevant information but will not provide training in changing thinking styles.
  Arms: Psychoeducation with treatment as usual

SUMMARY:
This study will conduct a randomized controlled trial of Cognitive Bias Modification for Interpretation (CBM-I) as an augmentation to treatment as usual for obsessive compulsive disorder (OCD). CBM-I is a digital intervention designed to directly manipulate interpretation bias through repeated practice on a training task, thereby inducing cognitive changes in a relatively automatic or implicit manner. Specifically, this study will examine the feasibility, acceptability, and clinical outcomes associated with CBM-I.

Adults with obsessive compulsive disorder (OCD) will be recruited from a treatment program for this disorder and participants will be randomly assigned to either receive: 1) up to 12 sessions of CBM-I, or or up to 12 sessions of psychoeducation as a control condition.

ELIGIBILITY:
Inclusion Criteria:

* 1) OCD Institute patients
* 2) adults (> 18 years old)
* 3) able to complete a computer task for 20 minutes
* 4) consent to main OCD Institute study protocol
* 5) primary diagnosis of OCD (as measured by a score of >16 on the Y-BOCS and a clinical diagnosis of OCD by their treatment team
* 6) score of >131 on the Obsessive Beliefs Questionnaire-44 at admission [which is 1 SD above the mean score of the non-clinical sample reported in the original validation paper by the Obsessive Compulsive Cognitions Working Group (2005)]

Exclusion Criteria:

* 1) Currently experiencing acute symptoms of psychosis
* 2) Psychotic disorder diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Average Score on Yale-Brown Obsessive Compulsive Scale | Weeks 0, 4, and 8
  Interviewer-rated measure of OCD symptoms. It is 19 items, with only items 1-10 scored (from 0-4). Total scores range from 0-40, with higher scores reflecting greater severity.

SECONDARY OUTCOMES:
Change in Average Score on Obsessive Beliefs Questionnaire | Time Frame: Weeks 0, 2, 4, and 8
  Measure of interpretation biases, specifically: Inflated Responsibility/Overestimation of Threat, Perfectionism/Intolerance of Uncertainty, and Importance/Control of Thoughts. 44-item self-report measure, items scored 1-7 and summed; greater scores indicate greater severity.

CONTACTS AND LOCATIONS:
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States